CLINICAL TRIAL: NCT04539808
Title: NeoOPTIMIZE: An Open-Label, Phase II Trial to Assess the Efficacy of Adaptive Switching of FOLFIRINOX or Gemcitabine/Nab-Paclitaxel as a Neoadjuvant Strategy for Patients With Resectable and Borderline Resectable/Locally Advanced Unresectable Pancreatic Cancer
Brief Title: NeoOPTIMIZE: Early Switching of mFOLFIRINOX or Gemcitabine/Nab-Paclitaxel Before Surgery for the Treatment of Resectable, Borderline Resectable, or Locally-Advanced Unresectable Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Charles D Lopez, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00021614; NCI-2020-06277 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00021614 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Adenocarcinoma; Stage 0 Pancreatic Cancer American Joint Committee on Cancer v8; Stage I Pancreatic Cancer American Joint Committee on Cancer v8; Stage III Pancreatic Cancer American Joint Committee on Cancer v8; Stage IV Pancreatic Cancer American Joint Committee on Cancer v8
MeSH Terms: interventions — Capecitabine; Fluorouracil; dehydroftorafur; Irinotecan; Leucovorin; Losartan; Oxaliplatin; Radiotherapy; Radiation; X-Rays; Specimen Handling; Gemcitabine; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (mFOLFIRINOX, chemotherapy) (Experimental): mFOLFIRINOX REGIMEN: Oxaliplatin intravenously (IV) over 2 hrs, leucovorin calcium IV over 2 hrs, and irinotecan hydrochloride IV over 90 minutes on day 1. Also receive fluorouracil IV over 46 hrs starting on day 1. Repeats every 14 days for up to 4 cycles. Those with response and no disease progression may receive an additional 2 months.
  GA REGIMEN: Those with disease progression or toxicity to mFOLFIRINOX switch to GA regimen comprising gemcitabine hydrochloride IV over 30-60 mins and nab-paclitaxel IV over 30-40 mins on days 1, 8, and 15. Repeats every 28 days for 2 cycles.
  LOSARTAN: Cycle 1 day 1, start losartan potassium orally once daily until end of RT.
  RT/SURGERY: Short-course RT for 10 fractions over 5 days weekly or long-course RT with 15-25 fractions over 5 days weekly along with oral capecitabine twice daily on Monday-Friday or fluorouracil IV over 5-7 days weekly until completion of RT. Patients then undergo surgery 1-4 weeks following RT
  Interventions: Drug: Capecitabine; Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Drug: Leucovorin Calcium; Drug: Losartan Potassium; Drug: Oxaliplatin; Radiation: Radiation Therapy; Procedure: Resection; Procedure: Diagnostic Imaging; Procedure: Biospecimen Collection; Drug: Gemcitabine; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U-101440E
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Losartan Potassium — Given PO
  Other Names: Cozaar; losartan
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Radiation: Radiation Therapy — Undergo short-course or long-course RT
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection
Procedure: Diagnostic Imaging — Undergo diagnostic imaging
  Other Names: Medical Imaging
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Gemcitabine — Given IV
  Other Names: Gemcitabine hydrochloride; Gemzar
Drug: Nab paclitaxel — Given IV
  Other Names: Albumin-bound paclitaxel; Protein-bound paclitaxel; Abraxane

SUMMARY:
This phase II trial evaluates whether early switching from modified fluorouracil/irinotecan/leucovorin/oxaliplatin (mFOLFIRINOX) chemotherapy regimen to a combination of gemcitabine and nab-paclitaxel (GA) before surgery is effective in treating patients with pancreatic cancer that can be surgically removed (resectable or borderline resectable), or that has spread to nearby tissue or lymph nodes and cannot be removed by surgery (locally-advanced unresectable). Chemotherapy drugs, such as fluorouracil, irinotecan, leucovorin, oxaliplatin, gemcitabine, and nab-paclitaxel work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. The study will also evaluate the drug losartan in combination with mFOLFIRINOX or GA.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the rate of margin-negative (R0) resection in participants with resectable or borderline resectable pancreatic cancer (BRPC) following treatment using NeoOPTIMIZE adaptive therapy (i.e., FOLFIRINOX alone, or switch to GA).

SECONDARY OBJECTIVES:

I. To determine the progression-free survival (PFS) of resectable or BRPC participants that received NeoOPTIMIZE adaptive therapy (i.e., FOLFIRINOX, or switch to GA).

II. To determine the PFS for the subset of resectable or BRPC participants that received NeoOPTIMIZE adaptive therapy, plus preoperative radiation therapy (RT).

III. To determine the disease-free survival (DFS) of resectable or BRPC participants that received NeoOPTIMIZE adaptive therapy (i.e., FOLFIRINOX, or switch to GA).

IV. To determine the DFS for the subset of resectable or BRPC participants that received NeoOPTIMIZE adaptive therapy plus preoperative RT.

V. To determine the overall survival (OS) of resectable or BRPC participants that received NeoOPTIMIZE adaptive therapy.

VI. To determine the OS for the subset of resectable or BRPC participants that received NeoOPTIMIZE adaptive therapy plus preoperative RT.

VII. To assess the surgical complications of resectable or BRPC participants that undergo surgical resection.

VIII. To assess 30-day post-operative mortality of participants with resectable or BRPC that undergo surgical resection.

IX. To assess safety of NeoOPTIMIZE adaptive therapy (all participants).

EXPLORATORY OBJECTIVES:

I. To monitor changes in CA19-9 levels (all participants). II. To determine the rate of margin-negative (R0) resection in patients with locally advanced pancreatic cancer (LAPC), following treatment using NeoOPTIMIZE adaptive therapy (i.e., FOLFIRINOX alone, or switch to GA).

III. To determine the PFS of LAPC participants that received NeoOPTIMIZE adaptive therapy (i.e., FOLFIRINOX, or switch to GA).

IV. To determine the PFS for the subset of LAPC participants that received NeoOPTIMIZE adaptive therapy plus preoperative radiation therapy (RT).

V. To determine the disease-free survival (DFS) of LAPC participants that received NeoOPTIMIZE adaptive therapy (i.e., FOLFIRINOX, or switch to GA).

VI. To determine the DFS for the subset of LAPC participants that received NeoOPTIMIZE adaptive therapy plus preoperative RT.

VII. To determine the OS of LAPC participants that received NeoOPTIMIZE adaptive therapy.

VIII. To determine the OS for the subset of LAPC participants that received NeoOPTIMIZE adaptive therapy plus preoperative RT.

IX. To assess the surgical complications of LAPC participants that undergo surgical resection.

X. To assess 30-day post-operative mortality of LAPC participants who undergo surgical resection.

OUTLINE:

mFOLFIRINOX REGIMEN: Patients receive oxaliplatin intravenously (IV) over 2 hours, leucovorin calcium IV over 2 hours, and irinotecan hydrochloride IV over 90 minutes on day 1. Patients also receive fluorouracil IV over 46 hours starting on day 1. Treatment with mFOLFIRINOX repeats every 14 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo disease restaging (re-stage I). Patients with radiographic response and no disease progression receive mFOLFIRINOX for an additional 2 months (approximately 4 cycles). Patients then undergo second re-staging (re-stage II).

GA REGIMEN: After re-stage I, patients with disease progression or toxicity to mFOLFIRINOX (per assessment of the treating physician) switch to receive the GA regimen comprising gemcitabine hydrochloride IV over 30-60 minutes and nab-paclitaxel IV over 30-40 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo second re-staging (re-stage II). Patients may be switched to GA regimen from FOLFIRINOX regimen prior to re-stage I (per assessment of the treating physician).

LOSARTAN: Starting cycle 1 day 1, patients also receive losartan potassium orally (PO) once daily (QD) until completion of RT in the absence of disease progression or unacceptable toxicity.

RT/SURGERY: Patients with no vascular tumor involvement at re-stage II, undergo surgery 1-4 after completion of chemotherapy. Patients with resolution of tumor contact with pancreatic vasculature at re-stage II, undergo short-course RT to receive a total of 10 fractions over 5 days weekly (Monday-Friday). Patients with tumor vessel involvement that is persistent at re-stage II, undergo long-course RT to receive a total of 15-25 fractions over 5 days weekly (Monday-Friday), and receive capecitabine PO twice daily (BID) on Monday-Friday or fluorouracil IV over 5-7 days weekly until completion of RT. Patients then undergo surgery 1-4 weeks after completion RT.

Patients undergo diagnostic imaging as clinically indicated throughout the trial. Patients also undergo blood sample collection throughout the trial.

After completion of study treatment, patients are followed up as clinically indicated and following institutional standards, and then every 3 months for 6 months, and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Cytologic or histologic proof pancreatic ductal carcinoma is required prior to study entry

  * If a biopsy (e.g., endoscopic ultrasound [EUS]-guided fine needle aspiration [FNA]) is planned per standard of care, the participant may be asked to consent to the additional collection of tumor tissue for research
* No evidence of metastatic disease as determined by chest computed tomography (CT) scan, abdomen/pelvis computed tomography (CT) scan (or magnetic resonance imaging [MRI] with gadolinium and/or manganese) within the 45-day window of study entry or prior to the one cycle of standard of care (SOC) administered before study entry, which is consistent with the standard of care

  * Note: On a case by case basis, for participants who enroll on trial after having received up to 1 month of standard of care chemotherapy per Investigator discretion, baseline radiographic imaging performed per institutional guidelines prior to SOC chemotherapy treatment may be used per investigator discretion to fulfill baseline radiographic imaging criteria even if performed > 45 days prior to official study entry.
* Diagnostic staging laparoscopy is not required for study eligibility

  * If staging laparoscopy is planned per standard of care, the participant may be asked to consent to the collection of tumor tissue for research
* At time of screening, per National Comprehensive Cancer Network (NCCN) criteria, must have either:

  * Resectable pancreatic ductal adenocarcinoma (PDAC), defined as no arterial tumor contact (celiac axis [CA], superior mesenteric artery [SMA], or common hepatic artery [CHA]), or
  * Node positive disease as defined by CT, MRI, or EUS imaging, or
  * Borderline resectable PDAC, defined as:

    * For tumors of the head or uncinate process:

      * Solid tumor contact with the superior mesenteric vein (SMV) or portal vein of > 180 degrees with contour irregularity of the vein or thrombosis of the vein, but with suitable vessel proximal and distal to the site of involvement, allowing for safe and complete resection and vein reconstruction
      * Solid tumor contact with the inferior vena cava
      * Solid tumor contact with the common hepatic artery without extension to the celiac axis or hepatic artery bifurcation, allowing for safe and complete resection and reconstruction
      * Solid tumor contact with the SMA =< 180 degrees
      * Solid tumor contact with variable anatomy (e.g., accessory right hepatic artery, replaced right hepatic artery, replaced common hepatic artery, and the origin of replaced or accessory artery), and the presence and degree of tumor contact should be noted if present, as it may affect surgical planning
    * For tumors of the body/tail:

      * Solid tumor contact with the celiac axis of =< 180 degrees
      * Solid tumor contact with the celiac axis >180 degrees without involvement of the aorta and with an intact and uninvolved gastroduodenal artery, thereby permitting a modified Appleby procedure (although some members of the consensus committee preferred this criterion to be in the unresectable category)
  * Locally-advanced, unresectable disease as defined by NCCN guidelines as follows:

    * Tumors of the head with SMA >= 180 degrees, or any celiac abutment, unreconstractable SMV or portal occlusion, or aortic invasion or encasement
    * Tumors of the body with SMA or celiac encasement 180 degrees, unreconstractable SMV or portal occlusion, or aortic invasion
    * Tumors of the tail with SMA or celiac encasement >= 180 degrees
    * Irrespective of location, all tumors with evidence of nodal metastasis outside of the resection field that are considered unresectable
* Must be deemed fit to undergo planned curative resection as determined by institutional standards
* No history of previous chemotherapy for pancreatic cancer. At the discretion of the principal investigator (PI), patient that have received no more than 1 month of systemic chemotherapy (e.g., mFOLFIRINOX), per standard of care, for the treatment of their PDAC may be eligible to participate
* For participants who will get INV losartan, baseline systolic blood pressure (BP) > 100 mm Hg taken as the average of 3 blood pressure readings
* Hemoglobin > 9 g/dL with no blood transfusion within 28 days of starting treatment (prior to the one month of standard of care chemotherapy allowed by the protocol or within 4 weeks of screening)

  * Note: On a case by case basis, for participants who enroll on trial after having received up to 1 month of standard of care chemotherapy per Investigator discretion, labs prior to initiation of SOC chemotherapy treatment may be used per Investigator discretion to fulfill screening lab requirements even if performed > 4 weeks prior to official study entry and/or there are more recent labs available from during chemotherapy treatment
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L (> 1000 cells/mm^3) (prior to the one month of standard of care chemotherapy allowed by the protocol or within 4 weeks of screening)

  * Note: On a case by case basis, for participants who enroll on trial after having received up to 1 month of standard of care chemotherapy per Investigator discretion, labs prior to initiation of SOC chemotherapy treatment may be used per Investigator discretion to fulfill screening lab requirements even if performed > 4 weeks prior to official study entry and/or there are more recent labs available from during chemotherapy treatment
  * May be waived on a case-by-case basis for patient populations recognized to have normal baseline values below this level
* Platelet count >= 100 x 10^9/L (> 100,000 per mm^3) (at time of registration and within 4 weeks prior to initiating study therapy)
* Creatinine =< 1.5 mg/dL OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 30 mL/min/1.73 m^2 for participants with creatinine levels > 1.5 x institutional upper limit of normal (ULN) prior to the one month of standard of care chemotherapy allowed by the protocol or within 4 weeks of screening)

  * Note: On a case by case basis, for participants who enroll on trial after having received up to 1 month of standard of care chemotherapy per Investigator discretion, labs prior to initiation of SOC chemotherapy treatment may be used per Investigator discretion to fulfill screening lab requirements even if performed > 4 weeks prior to official study entry and/or there are more recent labs available from during chemotherapy treatment
  * Creatinine clearance should be calculated per institutional standard. For participants with a baseline calculated creatinine clearance below normal institutional laboratory values, a measured baseline creatinine clearance should be determined. Individuals with higher values felt to be consistent with inborn errors of metabolism will be considered on a case-by-case basis
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN); or =< 2 x ULN or 2 down-trending values for individuals who have undergone biliary stenting prior to the one month of standard of care chemotherapy allowed by the protocol or within 4 weeks of screening)

  * Note: On a case by case basis, for participants who enroll on trial after having received up to 1 month of standard of care chemotherapy per Investigator discretion, labs prior to initiation of SOC chemotherapy treatment may be used per Investigator discretion to fulfill screening lab requirements even if performed > 4 weeks prior to official study entry and/or there are more recent labs available from during chemotherapy treatment
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN, OR two consecutive down-trending values for individuals who have undergone biliary stenting prior to the one month of standard of care chemotherapy allowed by the protocol or within 4 weeks of screening)

  * Note: On a case by case basis, for participants who enroll on trial after having received up to 1 month of standard of care chemotherapy per Investigator discretion, labs prior to initiation of SOC chemotherapy treatment may be used per Investigator discretion to fulfill screening lab requirements even if performed > 4 weeks prior to official study entry and/or there are more recent labs available from during chemotherapy treatment
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to initiating study therapy. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female participants of childbearing potential agree to use adequate methods of contraception starting with the first dose of study therapy through 30 days after the last dose of study therapy

  * Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year without an alternative medical cause
* Male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through 30 days after the last dose of study therapy
* Male patients must use a condom during treatment when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male participant should also use a highly effective form of contraception if they are of childbearing potential
* Participants currently receiving an angiotensin-converting enzyme (ACE) inhibitor or angiotensin II receptor blocker (ARB) will remain eligible for study participation. In such cases, losartan will not be assigned as part of the study intervention. These participants will continue to receive their ACE inhibitor or ARB per standard-of-care. The ACE inhibitor or ARB type should be recorded as a concomitant medication (including dose and frequency)

Exclusion Criteria:

* History of previous chemotherapy (other than no more than one cycle of standard systemic chemotherapy), targeted/biologic therapy, or radiation therapy for the treatment of their PDAC
* Evidence of metastasis to distant organs (liver, peritoneum, lung, others)
* Any other active malignancy or prior history of malignancy with less than a 90% cure rate in the judgement of the investigators
* Medical co-morbidities that are deemed to make risk of surgery unacceptably high as determined by institutional standards
* Personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest. Patients with cardiovascular conditions that are well-controlled in the clinical judgement of the treating oncologist are eligible to participate
* Recent major surgery (excluding laparoscopy) within 4 weeks prior to starting study treatment. Minor surgery within 2 weeks of starting study treatment. Patients must be recovered from effects of surgery
* Concomitant use of other anti-cancer therapy (chemotherapy, immunotherapy, hormonal therapy [hormone replacement therapy is acceptable]), not otherwise allowed in this study. Note: participation in other trials for supportive cancer care (e.g., cancer-related cachexia) interventions is permitted per PI discretion.
* Participants with a history of hypersensitivity reactions to study agents or their excipients. In cases of losartan hypersensitivity, losartan will be omitted and patient may still be eligible to participate
* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 30 days after the last dose of trial therapy
* Psychiatric illness/social situations, or any condition that, in the opinion of the investigator, would: interfere with evaluation of study treatment or interpretation of participant safety or study results, or substantially increase risk of incurring adverse events (AEs), or compromise the ability of the patient to give written informed consent
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2027-01-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Charles D Lopez, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Neoadjuvant Switch PDAC: Experimental: Treatment (mFOLFIRINOX, chemotherapy) mFOLFIRINOX REGIMEN: Oxaliplatin intravenously (IV) over 2 hrs, leucovorin calcium IV over 2 hrs, and irinotecan hydrochloride IV over 90 minutes on day 1. Also receive fluorouracil IV over 46 hrs starting on day 1. Repeats every 14 days for up to 4 cycles. Those with response and no disease progression may receive an additional 2 months.
  GA REGIMEN: Those with disease progression or toxicity to mFOLFIRINOX switch to GA regimen comprising gemcitabine hydrochloride IV over 30-60 mins and nab-paclitaxel IV over 30-40 mins on days 1, 8, and 15. Repeats every 28 days for 2 cycles.
  LOSARTAN: Cycle 1 day 1, start losartan potassium orally once daily until end of RT.
  RT/SURGERY: Short-course RT for 10 fractions over 5 days weekly or long-course RT with 15-25 fractions over 5 days weekly along with oral capecitabine twice daily on Monday-Friday or fluorouracil IV over 5-7 days weekly until completion of RT. Patients then undergo surgery 1-4 weeks following RT
Period: Overall Study
Arm/Group | Neoadjuvant Switch PDAC
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Switch PDAC
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 33
  Black or African American | 1
  Native American-Indigenous or Alaska Native | 3
  Asian | 1
  Native Hawaiian or other Pacific Islander | 1
  Not Reported/Unknown | 3
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Resectable or BRPC Participants With R0 Resection
Description: Using the surgery analysis set, the proportion of resectable or BRPC participants with R0 resection will be estimated with exact 95% CI.
Time Frame: Up to time of surgery
Population: Per protocol, the surgery safety analysis set is a sub-set of the safety analysis set that includes all participants who undergo surgical resection of their pancreatic cancer
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Switch PDAC
Number analyzed (Participants) | 30
percentage of participants | 93.33 [77.9 to 99.2]

2. Secondary Outcome: Progression-free Survival (PFS) NeoOPTIMIZE
Description: Using the efficacy analysis set, the estimated distribution of the PFS will be plotted using Kaplan Meier curves and reported with median survival and 95% confidence intervals if available. When feasible, sub-group analyses for the different treatment regimens (i.e., gemcitabine/nab-paclitaxel [GA] or modified fluorouracil/irinotecan/leucovorin/oxaliplatin [mFOLFIRINOX] +/- radiation therapy [RT] [i.e., short- or long-course, or both RT modalities combined]) will be performed for PFS.
Time Frame: From the start of neoadjuvant therapy (day 1) to the time of tumor progression, or death due to any cause, assessed up to 24 months
Reporting Status: Not Posted

3. Secondary Outcome: PFSNeoOPTIMIZE + Pre-operative (Preop)-RT
Description: Using the efficacy analysis set, the estimated distribution of the PFS will be plotted using Kaplan Meier curves and reported with median survival and 95% confidence intervals if available. When feasible, sub-group analyses for the different treatment regimens (i.e., GA or mFOLFIRINOX +/- RT [i.e., short- or long-course, or both RT modalities combined]) will be performed for PFS.
Time Frame: as for outcome 2
Reporting Status: Not Posted

4. Secondary Outcome: Disease-free Survival (DFS) NeoOPTIMIZE
Description: Using the surgery analysis set, the estimated distribution of the DFS will be plotted using Kaplan Meier curves and reported with median survival and 95% confidence intervals if available. Using the efficacy analysis set, the estimated distribution of the DFS will be plotted using Kaplan Meier curves and reported with median survival and 95% confidence intervals if available. When feasible, sub-group analyses for the different treatment regimens (i.e., GA or mFOLFIRINOX +/- RT [i.e., short- or long-course, or both RT modalities combined]) will be performed for DFS.
Time Frame: From the date of surgery to the time of tumor progression, or death due to any cause, assessed up to 24 months
Reporting Status: Not Posted

5. Secondary Outcome: DFSNeoOPTIMIZE + Preop-RT
Description: Using the efficacy analysis set, the estimated distribution of the DFS will be plotted using Kaplan Meier curves and reported with median survival and 95% confidence intervals if available. When feasible, sub-group analyses for the different treatment regimens (i.e., GA or mFOLFIRINOX +/- RT [i.e., short- or long-course, or both RT modalities combined]) will be performed for DFS.
Time Frame: From the date of surgery to the time of tumor progression, or death due to any cause, assessed up to 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival (OS) NeoOPTIMIZE
Description: Using the efficacy analysis set, the estimated distribution of the OS will be plotted using Kaplan Meier curves and reported with median survival and 95% confidence intervals if available. Using the efficacy analysis set, the estimated distribution of the OS will be plotted using Kaplan Meier curves and reported with median survival and 95% confidence intervals if available. When feasible, sub-group analyses for the different treatment regimens (i.e., GA or mFOLFIRINOX +/- RT [i.e., short- or long-course, or both RT modalities combined]) will be performed for OS.
Time Frame: From the start of neoadjuvant therapy (day 1) to death due to disease, assessed up to 24 months
Reporting Status: Not Posted

7. Secondary Outcome: OSNeoOPTIMIZE + Preop-RT
Description: Using the efficacy analysis set, the estimated distribution of the OS will be plotted using Kaplan Meier curves and reported with median survival and 95% confidence intervals if available. When feasible, sub-group analyses for the different treatment regimens (i.e., GA or mFOLFIRINOX] +/- RT [i.e., short- or long-course, or both RT modalities combined]) will be performed for OS.
Time Frame: From the start of neoadjuvant therapy (day 1) to death due to disease, assessed up to 24 months
Reporting Status: Not Posted

8. Secondary Outcome: Proportion of Resectable or BRPC Participants With Peri- and Post-operative Complications [Per the Clavien-Dindo Classification System]
Description: Using the surgery analysis set, for resectable and BRPC participants, the proportion of participants with peri- and post-operative complications occurring within 30 days is estimated.
Time Frame: Up to 30 days after surgery
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Switch PDAC
Number analyzed (Participants) | 30
percentage of participants | 97 [83 to 100]

9. Secondary Outcome: Proportion of Resectable or BRPC Participants That Die Within 30 Days of Surgery
Description: The proportion of resectable or BRPC participants that die within 30 days of surgery
Time Frame: At 30 days post-surgery
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Neoadjuvant Switch PDAC
Number analyzed (Participants) | 30
percent of participants | 3.3 [0.1 to 17.2]

10. Secondary Outcome: Incidence of Grade >= 3 Toxicities
Description: The incidence of grade >= 3 toxicities per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 will be determined using the safety analysis set. The exact 95% confidence interval will be reported with the point estimate of toxicity rate.
Time Frame: Up to 90 days after last dose of protocol-directed therapy
Population: Per protocol, the safety analysis set includes all enrolled participants who received at least 1 dose of systemic chemotherapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Switch PDAC
Number analyzed (Participants) | 42
percentage of participants | 54.8 [38.7 to 70.2]

11. Other Pre Specified Outcome: CA19-9 Serum Levels (U/ml)
Description: Using the safety analysis set, the levels of CA19-9 will be descriptively reported (across all participants).
Time Frame: Baseline up to 24 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Proportion of LAPC Participants With R0 Resection
Description: Using the surgery analysis set, the proportion of LAPC participants with R0 resection will be estimated with exact 95% CI.
Time Frame: From the start of neoadjuvant therapy (day 1) to time of surgery
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Switch PDAC
Number analyzed (Participants) | 1
percentage of participants | 100 [2.5 to 100]

13. Other Pre Specified Outcome: PFSNeoOPTMIZE for LAPC Cohort
Description: Results will be qualitatively described when statistical measures are not feasible.
Time Frame: From the start of neoadjuvant therapy (day 1) to time of tumor progression, or death due to any cause (up to 24 months from start of study treatment)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: PFSNeoOPTMIZE + Preop-RT for LAPC Subset
Description: Results will be qualitatively described when statistical measures are not feasible.
Time Frame: as for outcome 13
Reporting Status: Not Posted

15. Other Pre Specified Outcome: DFSNeoOPTMIZE for LAPC Cohort
Description: Results will be qualitatively described when statistical measures are not feasible.
Time Frame: From date of surgery to time of tumor progression, or death due to any cause (up to 24 months from start of study treatment)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: DFSNeoOPTMIZE + Preop-RT for LAPC Subset
Description: Results will be qualitatively described when statistical measures are not feasible.
Time Frame: as for outcome 15
Reporting Status: Not Posted

17. Other Pre Specified Outcome: OSNeoOPTMIZE for LAPC Cohort
Description: Results will be qualitatively described when statistical measures are not feasible.
Time Frame: From the start of neoadjuvant therapy (day 1) to death due to any cause, assessed up to 24 months from start of study treatment
Reporting Status: Not Posted

18. Other Pre Specified Outcome: OSNeoOPTMIZE + Preop-RT for LAPC Subset
Description: Results will be qualitatively described when statistical measures are not feasible.
Time Frame: as for outcome 17
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Proportion of LAPC Participants With Peri- and Post-operative Complications
Description: Using the surgery analysis set, for LAPC participants, the proportion of participants with peri- and post-operative complications occurring within 30 days is estimated.
Time Frame: From date of surgery to within 30 days from date of surgery
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Switch PDAC
Number analyzed (Participants) | 1
percentage of participants | 100 [2.5 to 100]

20. Other Pre Specified Outcome: Proportion of LAPC Participants Who Die Within 30 Days of Surgery
Description: Results will be qualitatively described when statistical measures are not feasible.
Time Frame: From date of surgery to 30 days post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Switch PDAC
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from start of first dose of study treatment up to and including 30 days following the date of last dose of study treatment.
Description: The safety analysis set includes all enrolled participants who received at least 1 dose of systemic chemotherapy
Arm/Group | Neoadjuvant Switch PDAC
All-Cause Mortality (participants affected / at risk) | 21/42
Serious Adverse Events (participants affected / at risk) | 22/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Switch PDAC (N=42)
Atrial flutter (Cardiac disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1)
Biliary tract infection (Infections and infestations) | 2 (3)
Appendicitis (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Hepatic infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Switch PDAC (N=42)
Anemia (Blood and lymphatic system disorders) | 3 (6)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 33 (50)
Diarrhea (Gastrointestinal disorders) | 30 (39)
Vomiting (Gastrointestinal disorders) | 12 (14)
Abdominal pain (Gastrointestinal disorders) | 10 (11)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 7 (10)
Mucositis oral (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 6 (10)
Bloating (Gastrointestinal disorders) | 6 (8)
Dyspepsia (Gastrointestinal disorders) | 5 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Obstruction gastric (Gastrointestinal disorders) | 1 (2)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 26 (39)
Edema limbs (General disorders) | 5 (5)
Fever (General disorders) | 4 (5)
Chills (General disorders) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (3)
Flu like symptoms (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Paresthesia (General disorders) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (3)
Biliary tract infection (Infections and infestations) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (3)
Appendicitis (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Hepatic infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (9)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 10 (12)
Aspartate aminotransferase increased (Investigations) | 6 (6)
Alkaline phosphatase increased (Investigations) | 5 (6)
Alanine aminotransferase increased (Investigations) | 5 (5)
Blood bilirubin increased (Investigations) | 4 (5)
Platelet count decreased (Investigations) | 4 (5)
Weight loss (Investigations) | 3 (3)
Creatinine increased (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 13 (20)
Anorexia (Metabolism and nutrition disorders) | 7 (10)
Dehydration (Metabolism and nutrition disorders) | 7 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (5)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 4 (5)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Infusion related reaction (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 25 (34)
Dysgeusia (Nervous system disorders) | 12 (12)
Dizziness (Nervous system disorders) | 8 (9)
Paresthesia (Nervous system disorders) | 5 (6)
Nervous system disorders - Other, specify (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 4 (5)
Dysphagia (Nervous system disorders) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 9 (12)
Confusion (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (4)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (4)
Hypertension (Vascular disorders) | 1 (3)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT04539808/Prot_SAP_000.pdf